CLINICAL TRIAL: NCT04600297
Title: Clinical Evaluation of 3D Printed Resin Composite Posterior Fixed Dental Prosthesis: A Prospective Clinical Trial up to 3 Years
Brief Title: 3 Years Clinical Evaluation of 3D Printed Resin Composite Fixed Dental Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Saremco Dental AG (Industry)
Responsible Party: Principal Investigator, Mehmet Muzaffer Ateş, Prof.Dr., Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68869993-511.06-.E.150622
Record Dates: First submitted 2020-10-13; First posted 2020-10-23 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Composite Resins; Dental Prosthesis
Keywords: 3D printed fixed prosthesis; resin composite dental prosthesis

STUDY DESIGN:
Intervention Model Description: Cases of one missing posterior tooth to be restored with 3D printed resin composite posterior FDP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D printed resin composite posterior FDP (Experimental): Three units posterior fixed dental prosthesis made with 3D printed resin composite material
  Interventions: Device: ELS Even Stronger (3D Printed Resin Composite)

INTERVENTIONS:
Device: ELS Even Stronger (3D Printed Resin Composite) — Missing of one premolar cases will be restored using the 3D Printed resin composite (ELS Even Stronger, Saremco, Switzerland). The steps of the procedure: Preparation, scanning, colour determination, design of the restoration, printing the restoration, adjusting occlusion, finishing and polishing, cementation.

SUMMARY:
In recent years there is a rapid increase in the use of computer aided design and production. Two main types of materials are used in the production of indirect CAD/CAM restorations namely resin composite based and ceramic ones. Mechanical properties and esthetics of ceramic materials are superior to resin composites but the advantages of intraoral repair, easy adjustments and polish of resin materials are undeniable. Improvements of mechanical properties of resin-based materials resulted in the development of resin composite blocks.

3D printed restorations, which can be performed as chairside in one session can be manufactured in case of any broken / chipping / debonding cases, without the need for repeated impression making. This saves time for the patient and the clinician. By using these 3D resin-based composite materials in fixed partial dentures, intraoral repairs can be performed. In addition, the high costs of burs and possible damage to the CAD/CAM blocks used in ceramic milling are eliminated when restoration are manufactured in printers with the DLP technology.

The objective of this study was to evaluate the clinical outcome of 3D printed posterior resin composite FDP restorations up to 3 years.

DETAILED DESCRIPTION:
The study will be carried out as a prospective study, with assessment of the restorations after three year. The project includes 3-unit posterior fixed dental prosthesis (FDP) for 70 cases.

Patients participating in the investigation are going to be informed by the "Clinicians" on the background and risk of the investigation. Patients have to give their written consent to participate in the investigation.

The treatment procedure includes the following steps:

Preparation scanning, colour determination, design of the restoration, printing the restoration, adjusting occlusion, finishing and polishing and cementation of the FDP.

The control procedures:

Two weeks after cementation, baseline control will be performed according to USPHS and FDI 2. The restorations will be evaluated at 3 years recall.

ELIGIBILITY:
Inclusion Criteria:

* Need for a three-unit posterior FDP
* One missing tooth from the second premolar to the second molar where 1st molar is missing (pontic replacing 1st molar)
* Presence of opposing natural dentition (either intact or restored with intracoronal or extracoronal fixed restorations), and with a minimum of 20 teeth)
* Only FPD s with end abutments (No cantilever)
* Sufficient length of the clinical crown (>5 mm)
* No obvious untreated caries, dental health problems (regularly checked by a dentist)
* Good or moderate oral hygiene (plaque score of less than 30% in anterior region be-fore treatment)
* No untreated periodontal disease (only DPSI 1, 2)
* Abutment teeth are vital or endodontically treated with a sealed root filling to the apical region, and have to be without apical periodontitis for the past 6 months.
* Subjects had to be over the age of 18, be classified according to the American Society of Anesthesiologists (ASA) as ASA I or ASA II, present with good oral hygiene, and be free of periodontal disease (probing depth and attachment levels within normal limits, no furcation involvement, and no mobility)
* Subjects had to agree to keep the scheduled recall appointments for data collection and maintenance and plan to stay in the area for at least 3 years.

Exclusion Criteria:

* Patients suffering from general health impairment
* Considerable horizontal and/or vertical mobility of teeth: tooth mobility index score 2 or - Considerable periodontal disease without treatment (DPSI 3-, 3+ and 4)
* Endodontic treatment with extensive loss of tooth tissue
* Subjects who presented with severe wear facets and/or reported parafunctional activi-ties such as clenching or nocturnal bruxism
* Subjects who were restored with a removable partial dental prosthesis (RPDP), unless the RPDP replaced the tooth that was planned to be restored in the study
* Subjects who were pregnant during the duration of the study
* Subjects who are known to be allergic to the ingredients of resin materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Modified FDI (World Dental Federation) criteria for dental restoration assessment | 3 years
  The FDI (World Dental Federation) criteria for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010. The criteria were categorized into three groups: esthetic, functional and biological parameters. Each criterion can be expressed with five scores, three for acceptable and two for non-acceptable (one for reparable and one for replacement). The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome. Two independent evaluators will evaluate the restorations by using modified FDI criteria.

SECONDARY OUTCOMES:
Plaque accumulation according to the Silness & Löe (1964) Plaque Index | 3 years
  0 = No plaque in the gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent
Gingival Inflammation according to the Silness & Löe (1964) Gingival Index. | 3 years
  0 = Normal gingival.
  1. = Mild inflammation-slight change in colour, slight oedema. No bleeding on probing
  2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing.
  3. = Severe inflammation-marked redness and oedema. Ulceration. Tendency to spontaneous bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mutlu Özcan, Prof.Dr., Principal Investigator — University of Zurich
Locations (1):
- İstanbul Medipol University, School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rekow ED. Dental CAD/CAM systems: a 20-year success story. J Am Dent Assoc. 2006 Sep;137 Suppl:5S-6S. doi: 10.14219/jada.archive.2006.0396. No abstract available. PMID 16950931
- [Background] Miyazaki T, Hotta Y, Kunii J, Kuriyama S, Tamaki Y. A review of dental CAD/CAM: current status and future perspectives from 20 years of experience. Dent Mater J. 2009 Jan;28(1):44-56. doi: 10.4012/dmj.28.44. PMID 19280967
- [Background] Ruse ND, Sadoun MJ. Resin-composite blocks for dental CAD/CAM applications. J Dent Res. 2014 Dec;93(12):1232-4. doi: 10.1177/0022034514553976. Epub 2014 Oct 24. PMID 25344335
- [Background] Zimmermann M, Ender A, Egli G, Ozcan M, Mehl A. Fracture load of CAD/CAM-fabricated and 3D-printed composite crowns as a function of material thickness. Clin Oral Investig. 2019 Jun;23(6):2777-2784. doi: 10.1007/s00784-018-2717-2. Epub 2018 Oct 27. PMID 30368664
- [Background] Alharbi A, Ardu S, Bortolotto T, Krejci I. Stain susceptibility of composite and ceramic CAD/CAM blocks versus direct resin composites with different resinous matrices. Odontology. 2017 Apr;105(2):162-169. doi: 10.1007/s10266-016-0258-1. Epub 2016 Jul 25. PMID 27456684
- [Background] Kamonwanon P, Hirose N, Yamaguchi S, Sasaki JI, Kitagawa H, Kitagawa R, Thaweboon S, Srikhirin T, Imazato S. SiO2-nanocomposite film coating of CAD/CAM composite resin blocks improves surface hardness and reduces susceptibility to bacterial adhesion. Dent Mater J. 2017 Jan 31;36(1):88-94. doi: 10.4012/dmj.2016-135. Epub 2016 Dec 6. PMID 27928105
- [Background] Mitra SB, Wu D, Holmes BN. An application of nanotechnology in advanced dental materials. J Am Dent Assoc. 2003 Oct;134(10):1382-90. doi: 10.14219/jada.archive.2003.0054. PMID 14620019
- [Background] Deliperi S, Bardwell DN. Clinical evaluation of direct cuspal coverage with posterior composite resin restorations. J Esthet Restor Dent. 2006;18(5):256-65; discussion 266-7. doi: 10.1111/j.1708-8240.2006.00033.x. PMID 16987320
- [Background] Yesil ZD, Alapati S, Johnston W, Seghi RR. Evaluation of the wear resistance of new nanocomposite resin restorative materials. J Prosthet Dent. 2008 Jun;99(6):435-43. doi: 10.1016/S0022-3913(08)60105-5. PMID 18514665
- [Background] Zimmermann M, Koller C, Reymus M, Mehl A, Hickel R. Clinical Evaluation of Indirect Particle-Filled Composite Resin CAD/CAM Partial Crowns after 24 Months. J Prosthodont. 2018 Oct;27(8):694-699. doi: 10.1111/jopr.12582. Epub 2017 Apr 19. PMID 28422359
- [Background] Shembish FA, Tong H, Kaizer M, Janal MN, Thompson VP, Opdam NJ, Zhang Y. Fatigue resistance of CAD/CAM resin composite molar crowns. Dent Mater. 2016 Apr;32(4):499-509. doi: 10.1016/j.dental.2015.12.005. Epub 2016 Jan 8. PMID 26777092
- [Background] Schlichting LH, Maia HP, Baratieri LN, Magne P. Novel-design ultra-thin CAD/CAM composite resin and ceramic occlusal veneers for the treatment of severe dental erosion. J Prosthet Dent. 2011 Apr;105(4):217-26. doi: 10.1016/S0022-3913(11)60035-8. PMID 21458646
- [Background] Magne P, Schlichting LH, Maia HP, Baratieri LN. In vitro fatigue resistance of CAD/CAM composite resin and ceramic posterior occlusal veneers. J Prosthet Dent. 2010 Sep;104(3):149-57. doi: 10.1016/S0022-3913(10)60111-4. PMID 20813228
- [Background] Magne P, Stanley K, Schlichting LH. Modeling of ultrathin occlusal veneers. Dent Mater. 2012 Jul;28(7):777-82. doi: 10.1016/j.dental.2012.04.002. Epub 2012 May 9. PMID 22575740
- [Background] El-Damanhoury HM, Haj-Ali RN, Platt JA. Fracture resistance and microleakage of endocrowns utilizing three CAD-CAM blocks. Oper Dent. 2015 Mar-Apr;40(2):201-10. doi: 10.2341/13-143-L. Epub 2014 Sep 30. PMID 25268039
- [Derived] Hobbi P, Ordueri TM, Ozturk-Bozkurt F, Toz-Akalin T, Ates MM, Ozcan M. Assessing the performance of 3D-printed resin composite posterior fixed dental prostheses: A 3-year prospective clinical trial. J Dent. 2025 Sep;160:105887. doi: 10.1016/j.jdent.2025.105887. Epub 2025 Jun 7. PMID 40490049
- [Derived] Hobbi P, Ordueri TM, Ozturk-Bozkurt F, Toz-Akalin T, Ates M, Ozcan M. 3D-printed resin composite posterior fixed dental prosthesis: a prospective clinical trial up to 1 year. Front Dent Med. 2024 Jun 4;5:1390600. doi: 10.3389/fdmed.2024.1390600. eCollection 2024. PMID 39917685